CLINICAL TRIAL: NCT03615404
Title: A Phase 1 Trial of CMV RNA-Pulsed Dendritic Cells With Tetanus-Diphtheria Toxoid Vaccine in Pediatric Patients and Young Adults With WHO Grade IV Glioma, Recurrent Malignant Glioma, or Recurrent Medulloblastoma
Brief Title: Cytomegalovirus (CMV) RNA-Pulsed Dendritic Cells for Pediatric Patients and Young Adults With WHO Grade IV Glioma, Recurrent Malignant Glioma, or Recurrent Medulloblastoma
Acronym: ATTAC-P
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gary Archer Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Gary Archer Ph.D., Assistant Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00092868
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Glioblastoma; Malignant Glioma; Medulloblastoma Recurrent; Pediatric Glioblastoma Multiforme; Pediatric Brain Tumor, Recurrent; Pediatric Brain Tumor
Keywords: glioblastoma; medulloblastoma; glioma; pediatric; recurrent; newly diagnosed; Pro00092868; Landi
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Recurrence; Medulloblastoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Tetanus Toxoid; Diphtheria Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CMV-DCs with GM-CSF and Td (tetanus toxoid) (Experimental): CMV-DCs are autologous dendritic cells derived from peripheral blood mononuclear cells (PBMCs) loaded with ribonucleic acid (RNA) encoding the human CMV matrix protein pp65 as a fusion protein with the full-length LAMP protein (pp65-flLAMP) plus GM-CSF and Td vaccine as adjuvants.
  Interventions: Biological: CMV-DCs with GM-CSF; Biological: Td (tetanus toxoid)

INTERVENTIONS:
Biological: CMV-DCs with GM-CSF — CMV-DCs are autologous dendritic cells derived from PBMCs loaded with RNA encoding the human CMV matrix protein pp65 as a fusion protein with the full-length LAMP protein (pp65-flLAMP) plus GM-CSF.
  Other Names: pp65-flLAMP DC with GM-CSF
Biological: Td (tetanus toxoid) — Patients will receive preconditioning with Td in the right groin, and approximately 6-24 hours later, they will receive their first CMV-DC vaccination. Patients will also receive Td preconditioning approximately 6-24 hours prior to their 4th vaccine and subsequent vaccines, if any.
  Other Names: Tetanus and Diphtheria Toxoid

SUMMARY:
The purpose of this study is to determine the feasibility and safety of administering CMV RNA-pulsed dendritic cells (DCs), also known as CMV-DCs, to children and young adults up to 35 years old with nWHO Grade IV glioma, recurrent malignant glioma, or recurrent medulloblastoma. Evidence for efficacy will also be sought. This will be a phase 1 study evaluating CMV-DC administration with tetanus toxoid (Td) preconditioning and Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF) adjuvant in children and young adults up to 35 years old with WHO grade IV glioma, recurrent malignant glioma, or recurrent medulloblastoma. This safety study will enroll a maximum of 10 patients.

DETAILED DESCRIPTION:
Participants in this study will undergo a leukapheresis procedure in which blood is collected into a machine that removes white blood cells and then returns the remainder of the blood back to the individual. The white blood cells removed from the blood are used to make the participant's study vaccine. Newly diagnosed patients will undergo standard radiation therapy (RT) with or without temozolomide after leukapheresis. If a patient has been diagnosed with a Grade IV glioma or recurrence of either malignant glioma or medulloblastoma, the study doctor may recommend "bridge therapy" after leukapheresis. Bridge therapy is approved or standard therapy for the tumor intended to bridge the time without the study drugs, dose-intensified temozolomide (DI-TMZ) or CMV-DC vaccine. All participants will undergo a cycle of "dose-intensified" temozolomide. Participants will receive Td pre-conditioning given as a shot in the right leg, six to 24 hours before receiving their 1st vaccine, which is also given as shots in the legs. If more than one vaccine is made, vaccines #2 and #3 will occur at 2-week intervals after the 1st vaccine. After the 3rd vaccine, there will be 4 weeks between vaccines for as many vaccines as the study team can prepare from the participant's leukapheresis.

Please note data collection will continue to occur outside of the defined primary outcomes for 2 exploratory objectives- describing changes in T cell response to CMV-DC vaccination and describing overall and progression-free survival of patients enrolled on the study. The percent change in pp65-specific T cell responses will be calculated from a pre-chemotherapy baseline, post-chemotherapy baseline, 1 week after Vaccine #3, and 1 week after final vaccine. Progression-free survival is defined as the time between starting DI TMZ and disease progression. Patients will be followed for overall survival for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age requirements:

   1. ≤ 35 years for patients with grade IV glioma or recurrent World Health Organization (WHO) grade IV glioma
   2. 3-35 years old for patients with recurrent medulloblastoma
2. Newly diagnosed or recurrent WHO grade IV glioma, recurrent WHO grade III glioma, or recurrent medulloblastoma (multifocal/disseminated disease is eligible, at the discretion of the PI)
3. Patients with WHO grade IV glioma who received surgery and radiation are eligible even without recurrence or progression
4. Patients must have recovered from all previous treatments including chemotherapy, radiation therapy, surgery, and other immunotherapies, etc.

   a. If the patient was receiving bevacizumab at the time of enrollment, the treating oncologist has the discretion of administering and adjusting bevacizumab 10 mg/kg every 14 days. The rationale for continuing patients on bevacizumab is to prevent rebound cerebral edema commonly seen after stopping this agent.
5. Laboratory Studies:

   1. Platelets ≥ 100,000 cells/mm3
   2. Creatinine ≤ 1.2 x upper limit of normal (ULN)
   3. Total bilirubin, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), alkaline phosphatase ≤ 2.5 x ULN
   4. Neutrophil count ≥ 1000 cells/mm3
   5. Hemoglobin ≥ 9 g/dl prior to biopsy (can be transfused)
6. Able to undergo brain MRI with and without contrast
7. Karnofsky Performance Status (KPS) ≥ 70 or Lansky Performance Status (LPS) ≥ 70
8. A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients (if 18 years old or older) or their parent(s) or guardian(s) (if younger than 18 years old) must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study.
9. For females of childbearing potential, negative serum pregnancy test within 48 hours of leukapheresis
10. Females of childbearing potential must be willing to use acceptable contraceptive method to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug
11. Males with female partners of childbearing potential must agree to practice adequate contraceptive methods throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug
12. Newly diagnosed WHO grade IV glioma patients only: must be expected to complete standard of care radiation (minimum ~54 Gray)

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible)
2. Disease outside of the central nervous system (CNS)
3. Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C seropositive
4. Known active infection requiring intravenous (IV) antibiotics or active immunosuppressive disease
5. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization
   2. Transmural myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at initiation of Radiation Therapy (XRT)/Temozolomide (TMZ)
   4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at initiation of XRT/TMZ for newly diagnosed patients or at initiation of dose-intensified (DI) TMZ for recurrent patients
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive
   7. Patients with autoimmune disease requiring medical management with immunosuppressant(s)
   8. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
   9. Active connective tissue disorders such as lupus or scleroderma that, in the investigator's opinion, place the patient at high risk for radiation toxicity
6. Pregnant or lactating women
7. Prior allergy to TMZ, GM-CSF, gadolinium (Gd), or Td
8. Prior history of brachial neuritis or Guillain-Barré syndrome
9. Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry
10. Patients receiving > 0.1mg/kg or 4mg/day dexamethasone or equivalent

10. For recurrent patients only: Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used:

1. Patients who have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from the side effects of such therapy. If the patient was receiving bevacizumab at the time of enrollment, the treating oncologist has the discretion of administering and adjusting bevacizumab 10 mg/kg every 14 days.
2. Patients who have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from the side effects of such therapy

Ages: 0 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu
- See also: The Preston Robert Tisch Brain Tumor Center at Duke Pediatric Program — https://tischbraintumorcenter.duke.edu/pediatrics

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled at a single institution, Duke University Medical Center.
Pre-assignment Details: All patients were enrolled into one cohort; no randomization occurred.
Period: Overall Study
Arm/Group | CMV-DCs With GM-CSF and Td (Tetanus Toxoid)
Started | 11
Completed | 9
Not Completed | 2
Not completed — Death | 1
Not completed — vaccine did not pass quality assurance | 1

BASELINE CHARACTERISTICS:
Arm/Group | CMV-DCs With GM-CSF and Td (Tetanus Toxoid)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients for Whom 3 or More Vaccines Can be Made
Description: Percentage of patients for whom three or more vaccines can be generated from the pre-treatment leukapheresis
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CMV-DCs With GM-CSF and Td (Tetanus Toxoid)
Number analyzed (Participants) | 11
percentage of participants | 90.9 [58.7 to 99.8]

2. Primary Outcome: Percentage of Patients Who Experience Unacceptable Toxicity
Description: Percentage of patients who experience unacceptable toxicity from CMV-DC administration
Time Frame: 1 year
Population: One eligible patient had a leukapheresis (evaluable for feasibility), but was withdrawn from the study due to clinical decline prior to receiving any treatment (not evaluable for safety).
Measure: Number; unit: percentage of patients
Arm/Group | CMV-DCs With GM-CSF and Td (Tetanus Toxoid)
Number analyzed (Participants) | 10
percentage of patients | 0

ADVERSE EVENTS:
Time Frame: 2 years from study registration
Arm/Group | CMV-DCs With GM-CSF and Td (Tetanus Toxoid)
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMV-DCs With GM-CSF and Td (Tetanus Toxoid) (N=9)
Anemia (Blood and lymphatic system disorders) | 4
Sinus tachycardia (Cardiac disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Injection site reaction (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 1
Muscle weakness left-sided (Nervous system disorders) | 1
Muscle weakness right-sided (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03615404/Prot_SAP_000.pdf